CLINICAL TRIAL: NCT05715996
Title: Application of Mixed Reality Technique for Percutaneous Lung Nodule Localization: A Prospective, Randomized, Controlled Trial
Acronym: MR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xinghua Cheng, MD, Shanghai Chest Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ShanghaiChestMR
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer
Keywords: mixed reality; Localization; sublobectomy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mixed reality guided localization group (Experimental): Application of mixed reality technique for percutaneous lung nodule localization.
  Interventions: Device: mixed reality guided localization
- Computerized tomography (CT) guided localization group (No Intervention): Computerized tomography (CT) guided percutaneous lung nodule localization.

INTERVENTIONS:
Device: mixed reality guided localization — In this study, MR was utilized to assist in the localization of pulmonary nodule during sublobectomy lung resection in patient to assess the accuracy of the technique.
  Arms: mixed reality guided localization group

SUMMARY:
With the popularization of CT screening, the detection rate of small lung nodules has greatly increased. Therefore, the clinical thoracoscopic lung nodule biopsy and sub-lobectomy for radical resection of lung cancer are greatly required. Accurate resection of lung nodule depends on precise localization of pulmonary nodules. However, preoperative CT-guided Hook- wire positioning under local anesthesia, which is the current primary localization method, requires high equipment and expense, and may cause physical and mental trauma to the patient. Augmented reality (AR) is an innovative technology that superimpose a virtual scene into the real environment by fusing images, videos, or computer-generated models with patients during surgical operations. It can visually display the anatomical structures of organs or lesions, which significantly improves surgical efficiency. This project intends to use AR technology to localize the solitary pulmonary nodule (SPN) before surgery, compared with CT-guided Hook-wire localization. Compared with the localization of SPNs under CT guidance, AR-assisted localization technology apparently is less time-consuming and can be performed immediately before surgery under general anesthesia, lessening pain, reduce costs of time and equipment, increase the success rate of sub-lobectomy, and improve the overall efficiency of surgical treatment of pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18years of age;
2. There was no distant metastasis in preoperative clinical evaluation;
3. The attending physician evaluated and confirmed the need for lung nodule localization and sub-lobectomy;
4. Target lung nodule diameter ≤ 2cm
5. The inner edge of the target node is at least 2 cm from the pulmonary artery or pulmonary vein
6. preoperative ECOG physical state score 0/1;
7. Volunteer to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. More than two lung nodules need to be removed at the same time.
2. The target node is located in the scapular region. Because percutaneous localization is obstructed by the scapula, percutaneous localization of pulmonary nodules is not suitable for such patients.
3. The patient has uncontrollable mental illness and cannot make subjective assessment.
4. After being selected, severe complications (unable to tolerate surgery or anesthesia) occurred before operation are not suitable or the treatment plan of the study cannot be implemented as planned;
5. After being selected, the patient's condition changes and needs to be changed from elective surgery to emergency surgery after being confirmed by the competent doctor;
6. At any stage after entering the study, the patient voluntarily requests to withdraw or discontinue treatment due to personal reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy of nodule localization | 30 minutes
  The deviation between the local quantizer and the target nodule center was evaluated. The deviation is expressed as vertical deviation, anteroposterior deviation and horizontal deviation in three dimensions. The total deviation of nodule localization is calculated as the square root of the sum of squares of each dimension.

SECONDARY OUTCOMES:
Operation duration | 30 minutes
  Since the start/end point of CT-guided pulmonary nodule localization may be arbitrary and there may be differences between different researchers, the program duration is derived from the CT scanning parameters and calculated as the length of time between the initial scan and the final scan. The hybrid reality guided positioning time is automatically recorded by the system from the beginning of registration to the completion of positioning
Incidence of complications | 7 days
  Including pneumothorax, hemoptysis, circulation changes caused by bleeding, pleural reaction, etc
Radiation exposure dose | 30 minutes
  The dose length product (DLP) was used to quantify the total radiation received by patients during the localization of pulmonary nodules. In addition, after the scanning process, the DLP value is directly displayed on the screen of the CT scanner. In order to estimate the relative amount of radiation dose, the effective dose (ED) is also calculated according to the DLP value
Postoperative puncture pain assessment | 7 days
  On the first day after the operation, when the patient was fully awake, the pain degree of the patient during the positioning process was evaluated by using the NRS (digital scoring method) and the Digital Assessment Scale of Pain Degree. The degree of pain is expressed in 0-10 numbers, 0 means no pain, and 10 means the most severe pain. It is left to the patient to choose a number that best represents the degree of pain, and the medical staff will select the corresponding number according to the patient's description of pain. According to the corresponding number of pain, the pain degree is divided into mild pain (1-3), moderate pain (4-6), and severe pain (7-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Zuodong Song, Shanghai, Shanghai Municipality, China